CLINICAL TRIAL: NCT03387657
Title: A Phase 1, Single-Center, Open-Label, Two-Period, Single-Sequence, Multiple Dosing Drug-Drug Interaction Study of Sotagliflozin and Hydrochlorothiazide in Healthy Male and Female Subjects
Brief Title: A Drug to Drug Interaction Study of Sotagliflozin With Hydrochlorothiazide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT14905; U1111-1186-2718 (Other: UTN)
Record Dates: First submitted 2017-12-20; First posted 2018-01-02 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sotagliflozin + Hydrochlorothiazide (HCTZ) (Experimental): Sotagliflozin to be administered alone in Period 1. HCTZ to be given in Period 2 for 4 days followed immediately by HCTZ and sotagliflozin for 5 days.
  Interventions: Drug: Sotagliflozin (SAR439954); Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: Tablet
  Route of administration: Oral
Drug: Hydrochlorothiazide — Pharmaceutical form: Tablet
  Route of administration: Oral

SUMMARY:
Primary Objective:

To assess the effects of multiple-dose hydrochlorothiazide (HCTZ) on the steady-state pharmacokinetics (PK) of sotagliflozin.

Secondary Objectives:

* To assess the safety and tolerability of multiple-dose sotagliflozin with and without co-administration of multiple-dose HCTZ
* To assess the effects of multiple-dose sotagliflozin on the steady-state PK of HCTZ
* To assess the effects of multiple-dose HCTZ on the steady-state PK of sotagliflozin-3-O-glucuronide

DETAILED DESCRIPTION:
Duration of the study for each subject will be between 33 to 77 days, including screening up to 28 days, 5 days of treatment Period 1, washout period of 7-21 days, 9 days of treatment Period 2, and follow-up period of 10-14 days after last dose of the Investigational Medicinal Product (IMP) in Period 2.

ELIGIBILITY:
Inclusion criteria :

* Male or female subjects, between 18 and 55 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 30.0 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs, electrocardiogram, and laboratory parameters.
* Female subject must use a double contraception method including a highly effective method of birth control, except if she has undergone sterilization at least 3 months earlier or is postmenopausal. The accepted double contraception methods include the use of 1 of the following contraceptive options: (1) intrauterine device; (2) condom or diaphragm or cervical/vault cap, in addition to spermicide. Menopause is defined as being amenorrheic for at least 2 years with plasma follicle stimulating hormone level >30 IU. Hormonal contraception is NOT acceptable in this study.
* Male subject, whose partners are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, a double contraception method according to the following algorithm: (condom) plus (spermicide or intra-uterine device or hormonal contraceptive) from the inclusion up to 4 months after the last dosing.
* Male subject, whose partners are pregnant, must use, during sexual intercourse, a condom from the inclusion up to 4 months after the last dosing.
* Male subject has agreed not to donate sperm from the inclusion up to 4 months after the last dosing.

Exclusion criteria:

* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Positive result on urine drug screen or alcohol test.
* Any contra-indications to hydrochlorothiazide, according to the applicable labeling.
* Any history or presence of deep leg vein thrombosis or embolism or a recurrent or frequent appearance of deep leg vein thrombosis in first degree relatives (parents, siblings or children).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Assessment of PK parameter: AUCtau | Period 1, days 2 to 6
  Sotagliflozin without HCTZ: AUC to the end of the dosing period (AUCtau)
Assessment of PK parameter: AUCtau | Period 2, days 6 to 10
  Sotagliflozin with HCTZ: AUCtau

SECONDARY OUTCOMES:
Assessment of PK parameter: AUCtau | Period 2, days 4 to 5
  HCTZ without sotagliflozin: AUCtau
Assessment of PK parameter: AUCtau | Period 2, days 9 to 10
  HCTZ with sotagliflozin: AUCtau
Assessment of PK parameter: AUCtau | Period 1, days 2 to 6
  Sotagliflozin-3-O-glucuronide without HCTZ: AUCtau
Assessment of PK parameter: AUCtau | Period 2, days 6 to 10
  Sotagliflozin-3-O-glucuronide with HCTZ: AUCtau
Assessment of PK parameter: Cmax | Period 2, days 4 to 5
  HCTZ without sotagliflozin: Maximum plasma concentration (Cmax)
Assessment of PK parameter: Cmax | Period 2, days 9 to 10
  HCTZ with sotagliflozin: Cmax
Assessment of PK parameter: Cmax | Period 1, days 2 to 6
  Sotagliflozin-3-O-glucuronide without HCTZ: Cmax
Assessment of PK parameter: Cmax | Period 2, days 6 to 10
  Sotagliflozin-3-O-glucuronide with HCTZ: Cmax
Assessment of PK parameter: tmax | Period 2, days 4 to 5
  HCTZ without sotagliflozin: Time to reach Cmax (tmax)
Assessment of PK parameter: tmax | Period 2, days 9 to 10
  HCTZ with sotagliflozin: tmax
Assessment of PK parameter: tmax | Period 1, days 2 to 6
  Sotagliflozin-3-O-glucuronide without HCTZ: tmax
Assessment of PK parameter: tmax | Period 2, days 6 to 10
  Sotagliflozin-3-O-glucuronide with HCTZ: tmax
Assessment of PK parameter: Cmax | Period 1, days 2 to 6
  Sotagliflozin without HCTZ: Cmax
Assessment of PK parameter: Cmax | Period 2, days 6 to 10
  Sotagliflozin with HCTZ: Cmax
Assessment of PK parameter: tmax | Period 1, days 2 to 6
  Sotagliflozin without HCTZ: tmax
Assessment of PK parameter: tmax | Period 2, days 6 to 10
  Sotagliflozin with HCTZ: tmax

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 8400001, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org